CLINICAL TRIAL: NCT05055713
Title: The Effects of Endoscopy Combined With Partial Splenic Artery Embolization in the Treatment of Cirrhosis With Esophageal and Gastric Varices Complicated With Hyperplenism or Splenomegaly:A Randomized Controlled Study.
Brief Title: A Randomized Controlled Study on the Treatment of Cirrhosis Combined With Hypersplenism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20200925-Qilu
Record Dates: First submitted 2021-09-16; First posted 2021-09-24 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2021-09

CONDITIONS: Liver Cirrhosis; Esophageal and Gastric Varices; Hypersplenism
Keywords: Esophageal and Gastric Varices; Hypersplenism; Rebleeding; Partial splenic artery embolization; Endoscopic Variceal Ligation
MeSH Terms: conditions — Liver Cirrhosis; Esophageal and Gastric Varices; Hypersplenism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Secondary prevention-1 (Experimental): Endoscopic therapy+ beta blockers
  Interventions: Procedure: Endoscopic therapy+ beta blockers
- Secondary prevention-2 (Experimental): Endoscopic therapy+ PSE+beta blockers
  Interventions: Procedure: Endoscopic therapy+ PSE+beta blockers
- Primary prevention-1 (Experimental): Endoscopic therapy
  Interventions: Procedure: Endoscopic therapy
- Primary prevention-2 (Experimental): Endoscopic therapy+ PSE
  Interventions: Procedure: Endoscopic therapy+ PSE
- Acute bleeding-1 (Experimental): Endoscopic therapy+somatostatin
  Interventions: Procedure: Endoscopic therapy+Somatostatin
- Acute bleeding-2 (Experimental): Endoscopic therapy+PSE+somatostatin
  Interventions: Procedure: Endoscopic therapy+PSE+Somatostatin

INTERVENTIONS:
Procedure: Endoscopic therapy+ beta blockers — Endoscopic variceal ligation (EVL) is for the secondary prophylaxis of esophageal variceal hemorrhage,and Cyanoacrylate injection is for gastric varices (GV).A standard dose of NSBB (carvedilol) was applied to patients according to the Baveno VI recommendations if there were no contraindications.
  Arms: Secondary prevention-1
Procedure: Endoscopic therapy+ PSE+beta blockers — Endoscopic variceal ligation (EVL) is for the secondary prophylaxis of esophageal variceal hemorrhage,and Cyanoacrylate injection is for gastric varices (GV).A standard dose of NSBB (carvedilol) was applied to patients according to the Baveno VI recommendations if there were no contraindications.Partial splenic embolization (PSE) is one of the intra-arterial therapeutic approaches to embolize 60-80% splenic blood flow.
  Arms: Secondary prevention-2
Procedure: Endoscopic therapy — Endoscopic variceal ligation (EVL) is for the secondary prophylaxis of esophageal variceal hemorrhage,and Cyanoacrylate injection is for gastric varices (GV).
  Arms: Primary prevention-1
Procedure: Endoscopic therapy+ PSE — Endoscopic variceal ligation (EVL) is for the secondary prophylaxis of esophageal variceal hemorrhage,and Cyanoacrylate injection is for gastric varices (GV).Partial splenic embolization (PSE) is one of the intra-arterial therapeutic approaches to embolize 60-80% splenic blood flow.
  Arms: Primary prevention-2
Procedure: Endoscopic therapy+Somatostatin — The first dose of 250 was injected intravenously, followed by a continuous iv infusion of 250 for 3-5 days. Endoscopic variceal ligation (EVL) is for the acute bleeding of esophageal variceal hemorrhage,and Cyanoacrylate injection is for gastric varices (GV).
  Arms: Acute bleeding-1
Procedure: Endoscopic therapy+PSE+Somatostatin — The first dose of 250 was injected intravenously, followed by a continuous iv infusion of 250 for 3-5 days. Endoscopic variceal ligation (EVL) is for the acute bleeding of esophageal variceal hemorrhage,and Cyanoacrylate injection is for gastric varices (GV).Partial splenic embolization (PSE) is one of the intra-arterial therapeutic approaches to embolize 60-80% splenic blood flow.
  Arms: Acute bleeding-2

SUMMARY:
The purpose of this study was to compare the effects of partial splenic artery embolization combined with endoscopic treatment and endoscopic treatment alone on portal hypertension in cirrhosis with hyperplenism or splenomegaly in esophageal and gastric varices.

DETAILED DESCRIPTION:
Although there have been many consensus opinions on the treatment of cirrhosis patients with esophageal and gastric variceal hemorrhage, there is no standard to follow for the treatment of cirrhosis patients with esophageal and gastric variceal hemorrhage combined with hypersplenism or splenomegalism, and studies show that the patients with cirrhosis combined with severe hypersplenism account for about 33%. It has been reported that partial splenic artery embolization is effective in the treatment of hypersplenism or splenomegaly caused by portal hypertension in liver cirrhosis, but for liver cirrhosis with esophageal and gastric varices hemorrhage in port or spleen large combined at the same time of endoscopic treatment should joint partial splenic artery embolization treatment remains controversial.Therefore, it is urgent to further study the effect of partial splenic artery embolization combined with endoscopic therapy on cirrhosis with esophageal and gastric variceal hemorrhage combined with hyperspleenism or splenomegaly.

ELIGIBILITY:
Secondary prevention:

Inclusion Criteria:

* Patients aged between 18 and 75 years
* Patients who had recovered from an episode of VH or patients who had survived from acute VH and there was no bleeding for consecutive 5 days
* Patients with a diagnosis of liver cirrhosis and portal hypertension on clinical examination, laboratory test, and imaging or histological examination
* Patients with hypersplenism and thrombocytopenia (platelets < 100,000/µL).

Exclusion Criteria:

* Previous therapy (splenectomy, PSE, EVL, tissue adhesive injection, or usage of (NSBB) to prevent rebleeding
* Bleeding from isolated gastric or ectopic varices
* Hepatocellular carcinoma or other malignant tumors
* Contraindications for the use of NSBBs, hepatic failure, and Child-Pugh class C with large amount ascites, or grade 3-5 hepatic encephalopathy, or prothrombin activity ≤ 40%
* Hepatic failure
* Contraindications for PSE
* Pregnancy and lactation
* Inability to sign the informed consent.

Primary prevention:

Inclusion Criteria:

* Patients aged between 18 and 75 years
* Moderate to severe esophageal (and/or) gastric varices
* Patients with a diagnosis of liver cirrhosis and portal hypertension on clinical examination, laboratory test, and imaging or histological examination
* Patients with hypersplenism and thrombocytopenia (platelets < 100,000/µL).

Exclusion Criteria:

* Previous therapy (splenectomy, PSE, EVL, tissue adhesive injection, or usage of (NSBB) to prevent rebleeding
* Bleeding from isolated gastric or ectopic varices
* Hepatocellular carcinoma or other malignant tumors
* Contraindications for the use of NSBBs, hepatic failure, and Child-Pugh class C with large amount ascites, or grade 3-5 hepatic encephalopathy, or prothrombin activity ≤ 40%
* Hepatic failure
* Contraindications for PSE
* Pregnancy and lactation
* Inability to sign the informed consent.

Acute bleeding:

Inclusion Criteria:

* Patients aged between 18 and 75 years
* Acute esophageal (and/or) gastric varices rupture and bleed <5 days
* Patients with a diagnosis of liver cirrhosis and portal hypertension on clinical examination, laboratory test, and imaging or histological examination
* Patients with hypersplenism and thrombocytopenia (platelets < 100,000/µL).

Exclusion Criteria:

* Previous therapy (splenectomy, PSE, EVL, tissue adhesive injection, or usage of (NSBB) to prevent rebleeding
* Bleeding from isolated gastric or ectopic varices
* Hepatocellular carcinoma or other malignant tumors
* Contraindications for the use of NSBBs, hepatic failure, and Child-Pugh class C with large amount ascites, or grade 3-5 hepatic encephalopathy, or prothrombin activity ≤ 40%
* Hepatic failure
* Contraindications for PSE
* Pregnancy and lactation
* Inability to sign the informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2020-09-25 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
rebleeding | 2 to 30days
  the rate of rebleeding after endoscopic therapy

CONTACTS AND LOCATIONS:
Overall Officials: Yanjing Gao, PhD.MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital , Shandong University, Jinan, Shandong, China